CLINICAL TRIAL: NCT02570646
Title: QuitAdvisorDDS: A Point-of-Care Tobacco Cessation Tool for Dental Settings
Acronym: QA-DDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jamie Studts (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); University of Alabama at Birmingham (Other); The National Dental Practice-Based Research Network (Network); Health Decision Technologies, LLC (Other)
Responsible Party: Sponsor-Investigator, Jamie Studts, Principle investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-155-E; R44DE021327 (NIH)
Record Dates: First submitted 2015-10-03; First posted 2015-10-07 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- QA-DDS (Experimental): Patients will receive exposure to the QA-DDS tool from their dental care practitioner.
  Interventions: Behavioral: QA-DDS

INTERVENTIONS:
Behavioral: QA-DDS — QuitAdvisorDDS is a point-of-care software tool to facilitate implementation of evidence-based tobacco treatment interventions in dental care settings.
  Other Names: QuitAdvisorDDS

SUMMARY:
Using a single-arm trial design, this study will examine the feasibility and acceptability of evaluating QuitAdvisorDDS, a clinical decision support software application designed to facilitate implementation of evidence-based tobacco treatment interventions into the dental setting. The study will examine the feasibility and acceptability of evaluating the impact of the QuitAdvisorDDS tool on patient outcomes related to tobacco use and cessation attempts as well as provider knowledge, attitudes, and practices regarding tobacco treatment. Practitioners (dentists and hygienists) will complete surveys at baseline and follow-up, while patients will complete surveys at baseline and 1-month follow-up. An embedded substudy will also evaluate the feasibility and acceptability of collecting biospecimens (saliva) to serve as biochemical verification of smoking status.

ELIGIBILITY:
Inclusion Criteria:

* Receives dental care from a participating practitioner;
* Is age 18 or older;
* Self-reports tobacco use within the past month;
* Willing to comply with all study procedures and be available for the duration of the study;
* Willing to provide verbal informed consent;
* Has access to a telephone, and agrees to receive text messages, emails, or telephone calls related to the study. (The patient's preferred method of contact will be ascertained).
* Willing to be contacted on a regular basis by each of these entities: the practice;Regional Coordinators (RC) and/or University of Kentucky (UK) researchers; and
* Willing to provide contact information of one person living at a different address who will know the patient's whereabouts in the event the patient cannot be reached.

Exclusion Criteria:

* Psychiatric disability or mental illness judged by the practitioner to be clinically significant so as to preclude informed consent or compliance with procedures of study visits.
* Cognitive impairment judged by the practitioner to be significant so as to preclude informed consent or compliance with procedures of study visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2015-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Primary Patient Acceptability A: Rate of Patient Wanting Provider to Use QA-DDS | Immediately Post-Consultation up to 1 week
  80% of participating patients must indicate that they would want their dental practitioner to continue to use QA-DDS.
Primary Patient Acceptability B: Rate of Patient Wanting to Use QA-DDS Patient Portal | 1-Month Follow-Up
  80% of participating patients must indicate that they would want to continue to use the QA-DDS Patient Portal.
Primary Patient Feasibility A: Rate of Patient Completion of 1-Month Follow-Up Survey | 1-Month Follow-Up
  80% of the enrolled dental care patients must complete the 1-month follow-up survey with the 7-day point prevalence measure of self-reported smoking status.

SECONDARY OUTCOMES:
Secondary Patient Acceptability A: Average QA-DDS Satisfaction Ratings Among Patients on 0-10 Scale | Immediately Post-Consultation up to 1 week
  Average QA-DDS satisfaction ratings among enrolled dental patients must be 7 or greater on a 0-10 scale.
Secondary Patient Feasibility A: Rate of Patient Accrual by Study Practices | 4-Month Follow-Up
  75% of the study practices must recruit 10 eligible dental patients within a 4-month recruitment phase

OTHER OUTCOMES:
Tertiary Patient Acceptability A1: Number of Patients Who Visit QA-DDS Patient Portal | 1-Month Follow-Up
  To evaluate the acceptability of the QA-DDS Patient Portal among enrolled dental patients, the percentage of enrolled patients who make at least one visit to the Patient Portal will be monitored
Tertiary Patient Acceptability A2: Number of Visits to QA-DDS Patient Portal Per Patient | 1-Month Follow-Up
  To evaluate the acceptability of the QA-DDS Patient Portal among enrolled dental patients, the number of visits to the Patient Portal per patient will be monitored
Tertiary Patient Acceptability B: Rate of QA-DDS Text Messaging Support Service Use as Measured by Number of Patient Subscriptions | 1-Month Follow-Up
  To evaluate the acceptability of the QA-DDS Text Messaging Support Service, the percentage of enrolled patients who subscribe to the Text Messaging Support Service will be monitored.
Tertiary Patient Feasibility A: Rate of Missing Data for Tobacco Use Among Patients | 1-Month Follow-Up
  Self-reported measures of tobacco use and history at the follow-up assessment must have less than 10% missing data among responding dental patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie L Studts, PhD, Principal Investigator — Associate Professor, University of Kentucky College of Medicine
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

REFERENCES:
- [Derived] Holliday R, Hong B, McColl E, Livingstone-Banks J, Preshaw PM. Interventions for tobacco cessation delivered by dental professionals. Cochrane Database Syst Rev. 2021 Feb 19;2(2):CD005084. doi: 10.1002/14651858.CD005084.pub4. PMID 33605440